CLINICAL TRIAL: NCT05969795
Title: Comparison of Live Birth Rate (> 24 Weeks) in Natural Cycle (NC) Single Euploid Frozen Embryo Transfers (FET) With Versus Without Luteal Phase Support (LPS)
Brief Title: Comparison of Live Birth Rate in Natural Cycle Single Euploid FET Versus Without Luteal Phase Support
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2306-ABU-009-BL
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Related; Infertility, Female
Keywords: implantation rate; infertility; pregnancy rate; natural cycle; luteal phase support; live birth; progesterone
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Progesterone; Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Other): Intermittent ultrasound scans to monitor follicular growth and serial measurements of serum LH, E2 and P4 levels throughout the cycle to determine ovulation. Embryo transfer (ET) will be scheduled on the fifth day after ovulation. Blood for P4 measurement will be drawn upon admission to the clinic for the ET procedure. P4 will be measured on day 5 or day 6 after the ET procedure and together with the hCG 10 days after ET procedure.
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Serial serum LH, E2, P4; Diagnostic Test: Serum P4 day of ET - Study Group; Procedure: Embryo transfer; Diagnostic Test: Serum hCG 10 days after ET; Diagnostic Test: Serum P4 10 days after ET
- Control Group (Other): Intermittent ultrasound scans to monitor follicular growth and serial measurements of serum LH, E2 and P4 levels throughout the cycle to determine ovulation. Embryo transfer (ET) will be scheduled on the fifth day after ovulation. Administer on FET day 200 mg of P4 and increase to 300 mg/day from the day after the ET onwards until the pregnancy test. Blood for P4 measurement will be drawn before starting LPS in form of vaginal progesterone. P4 will be measured on day 5 or day 6 after the ET procedure and together with the hCG 10 days after ET procedure. In case of an implantation, vaginal P4 will be continued until 7 weeks of pregnancy.
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Serial serum LH, E2, P4; Drug: Progesterone 100 Mg Vaginal Insert; Diagnostic Test: Serum P4 day of ET - Control Group; Procedure: Embryo transfer; Diagnostic Test: Serum hCG 10 days after ET; Diagnostic Test: Serum P4 10 days after ET

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — Intermittent transvaginal ultrasound throughout the cycle to monitor follicular growth
Diagnostic Test: Serial serum LH, E2, P4 — Serial measurements of serum Luteinizing Hormone (LH), Estradiol (E2) and Progesterone (P4 )levels throughout the cycle to determine ovulation. LH-surge is identified when a rise of 180% above the previous level occurred and ovulation is confirmed with a decrease in E2 concentration, and a rise of progesterone level to ≥ 1.0 ng/ml (Irani et al., 2017).
Drug: Progesterone 100 Mg Vaginal Insert — On day of ET procedure, to administer 200 mg of vaginal progesterone and increase to 300 mg/day from the day after the ET onwards until the pregnancy test. In case of an implantation, vaginal P4 will be continued until 7 weeks of pregnancy
  Other Names: Progesterone 100Mg Vag Tab
  Arms: Control Group
Diagnostic Test: Serum P4 day of ET - Control Group — Serum P4 will be drawn before starting LPS in form of vaginal progesterone on the day of ET procedure
  Arms: Control Group
Diagnostic Test: Serum P4 day of ET - Study Group — Serum P4 will be drawn when study group participants are admitted to the clinic for the ET procedure.
  Arms: Study Group
Procedure: Embryo transfer — The procedure in which embryo is placed in the uterus.
  Other Names: ET
Diagnostic Test: Serum hCG 10 days after ET — Pregnancy will be confirmed / excluded by measurement of serum hCG 10 days after ET procedure and a level of > 15 IU will be regarded as positive result. The definitions of biochemical, ectopic, clinical and ongoing pregnancy follow the ICMART criteria (Zegers-Hochschild, 2006)
Diagnostic Test: Serum P4 10 days after ET — Serum P4 will be drawn on day 5 or day 6 after the ET procedure and together with the hCG 10 days after ET procedure

SUMMARY:
To evaluate whether single euploid embryo transfer in NC without routinely administered LPS is non-inferior to NC with routinely administered LPS.

DETAILED DESCRIPTION:
In case the study will show that the live birth rate in single euploid NC frozen embryo transfer cycles without LPS is not inferior to NC cycles with LPS, treatment can be simplified, and participants comfort can be increased.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 40 years
* Regular ovulatory cycles
* Availability of at least one euploid embryo after Trophectoderm biopsy for PGT-A on day 5 or day 6
* Detection of ovulation by P4 rise > 1.0 ng/ml after LH surge
* P4 value of at least 5 ng/ml on day 4 after ovulation

Exclusion Criteria:

* History of repeated pre-menstrual spotting
* Factors affecting the implantation through anatomical changes of the uterus / ovaries or the tubes (adenomyosis, Asherman syndrome, endometriosis, uterine fibroids / polyps, isthmocele with intracavitary fluid presence, hydrosalpinx….)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 342 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 2 months
  Number of embryos which have produced ultrasonographic evidence of an intrauterine gestational sac per the total number of embryos transferred into the uterine cavity (Zegers-Hochschild et al., 2009).
Clinical pregnancy rate | 2 months
  hCG > 15 Iu/ml and ultrasound confirmation of a gestational sac
Live birth rate | 41 weeks
  Number of deliveries that resulted in a live born neonate, expressed per 100 embryo transfers (Zegers-Hochschild et al., 2009)
Serum P4 levels on ET day | 1 day
  Progesterone level on the day of embryo transfer
Serum E2 and P4 levels on day 5 or 6 after ET procedure | 6 days
  Estradiol and Progesterone levels on day 5 or 6 after embryo transfer
Serum E2 and P4 levels on day 10 after ET procedure | 10 days
  Estradiol and Progesterone levels on day 10 after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (3):
- United Arab Emirates (3):
  - ART Fertility Clinics LLC, Abu Dhabi
  - ART Fertility Clinics Al Ain, Al Ain City
  - ART Fertility Clinics Dubai, Dubai

REFERENCES:
- [Background] Bortoletto P, Prabhu M, Baker VL. Association between programmed frozen embryo transfer and hypertensive disorders of pregnancy. Fertil Steril. 2022 Nov;118(5):839-848. doi: 10.1016/j.fertnstert.2022.07.025. Epub 2022 Sep 25. PMID 36171152
- [Background] Csapo AI, Pulkkinen M. Indispensability of the human corpus luteum in the maintenance of early pregnancy. Luteectomy evidence. Obstet Gynecol Surv. 1978 Feb;33(2):69-81. doi: 10.1097/00006254-197802000-00001. No abstract available. PMID 341008
- [Background] Filicori M, Butler JP, Crowley WF Jr. Neuroendocrine regulation of the corpus luteum in the human. Evidence for pulsatile progesterone secretion. J Clin Invest. 1984 Jun;73(6):1638-47. doi: 10.1172/JCI111370. PMID 6427277
- [Background] Ginstrom Ernstad E, Wennerholm UB, Khatibi A, Petzold M, Bergh C. Neonatal and maternal outcome after frozen embryo transfer: Increased risks in programmed cycles. Am J Obstet Gynecol. 2019 Aug;221(2):126.e1-126.e18. doi: 10.1016/j.ajog.2019.03.010. Epub 2019 Mar 22. PMID 30910545
- [Background] Pape J, Levy J, von Wolff M. Early pregnancy complications after frozen-thawed embryo transfer in different cycle regimens: A retrospective cohort study. Eur J Obstet Gynecol Reprod Biol. 2022 Dec;279:102-106. doi: 10.1016/j.ejogrb.2022.10.015. Epub 2022 Oct 21. PMID 36308939
- [Background] Roelens C, Blockeel C. Impact of different endometrial preparation protocols before frozen embryo transfer on pregnancy outcomes: a review. Fertil Steril. 2022 Nov;118(5):820-827. doi: 10.1016/j.fertnstert.2022.09.003. PMID 36273850
- [Background] Soules MR, Clifton DK, Steiner RA, Cohen NL, Bremner WJ. The corpus luteum: determinants of progesterone secretion in the normal menstrual cycle. Obstet Gynecol. 1988 May;71(5):659-66. PMID 3357651
- [Background] Su S, Zeng M, Duan J. Luteal phase support for natural cycle frozen embryo transfer: a meta-analysis. Gynecol Endocrinol. 2022 Feb;38(2):116-123. doi: 10.1080/09513590.2021.1998438. Epub 2021 Nov 3. PMID 34730071
- [Background] Practice Committee of the American Society for Reproductive Medicine. The clinical relevance of luteal phase deficiency: a committee opinion. Fertil Steril. 2012 Nov;98(5):1112-7. doi: 10.1016/j.fertnstert.2012.06.050. Epub 2012 Jul 20. PMID 22819186
- [Background] von Versen-Hoynck F, Schaub AM, Chi YY, Chiu KH, Liu J, Lingis M, Stan Williams R, Rhoton-Vlasak A, Nichols WW, Fleischmann RR, Zhang W, Winn VD, Segal MS, Conrad KP, Baker VL. Increased Preeclampsia Risk and Reduced Aortic Compliance With In Vitro Fertilization Cycles in the Absence of a Corpus Luteum. Hypertension. 2019 Mar;73(3):640-649. doi: 10.1161/HYPERTENSIONAHA.118.12043. PMID 30636552
- See also: Shapiro BS, Garner FC, Aguirre M. The Freeze-All Cycle: A New Paradigm Shift in ART. In Nagy ZP, Varghese AC, Agarwal A, editors. In Vitro Fertilization [Internet] 2019;, p. 765-778. Springer International Publishing — http://link.springer.com/10.1007/978-3-319-43011-9_63